CLINICAL TRIAL: NCT04543929
Title: Effects of Innovative Aerobic Exercise Training in Cystic Fibrosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Principal Investigator, Dave Burnett, Ph.D., Chair Dept. of Respiratory Care and Diagnostic Science, University of Kansas Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00143513
Record Dates: First submitted 2020-09-02; First posted 2020-09-10 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-08

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- exercise (Active Comparator): exercise prescription + standard of care
  Interventions: Behavioral: exercise
- no exercise (No Intervention): no exercise prescription + standard of care

INTERVENTIONS:
Behavioral: exercise — partially supervised and home-based exercise activity
  Arms: exercise

SUMMARY:
The main objective of this study is to compare the effectiveness of two different exercise interventions in a patient-centered, home-based exercise program for improving cardiorespiratory-fitness in people with cystic fibrosis (CF). We hypothesize cystic fibrosis patients participating in a high intensity interval training (HIIT) group will experience greater improvements in cardiorespiratory-fitness than those in a moderate continuous training (MCT) group. Further, we plan to investigate the efficacy of the comparators on patient-centered outcomes.

DETAILED DESCRIPTION:
This study is a randomized control trial that compares MCT to HIIT using a patient-centered and home-based delivery model with CF Care Centers in the United States. Participants will be randomly allocated to either an MCT or HIIT arm. Both the MCT and HIIT interventions are accepted forms of prescribed exercise in clinical practice. The interventions will be delivered with a telehealth platform using internet (HIPAA-Compliant video), phone, and email/text support. All study sites will receive initial and on-going training and program facilitation to assure consistency of delivering the intervention. All participants across both arms visit their respective CF clinics on a regular basis for routine CF care. Thus, our research team will be able to coordinate all testing/assessment visits, including long-term (18-month timepoint), with participants throughout the study. The primary and secondary outcomes include important patient-centered outcomes as selected by our study's CF Patient and Stakeholder Advisory Board.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with Cystic Fibrosis
* Prescribed and taking for 28 days ivacaftor-tezacaftor-elexacaftor (Trikafta)
* 18 years and older

Exclusion Criteria:

* 17 years of age or less
* not eligible for ivacaftor-tezacaftor-elexacaftor (Trikafta)
* inability to exercise
* pregnancy
* status post lung transplantation
* already participating in more than 150 minutes of aerobic exercise per week

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2020-02-11 (Actual); Primary Completion 2020-06-23 (Actual); Study Completion 2020-06-23 (Actual)

PRIMARY OUTCOMES:
Aerobic Exercise Capacity - V02max | 18 months
  anaerobic threshold (V02max) measured via Sub-maximal cardiopulmonary exercise test (CPET)

SECONDARY OUTCOMES:
Pulmonary function testing | 18 months
  Standardized testing to measure forced expiratory volume 1 sec (FEV1)
Quality of Life measured by Cystic Fibrosis Questionnaire - Revised (CFQ-R) | 18 months
  cystic fibrosis questionnaire (CFQ-R) score. Standardized scores ranging from 0 to 100; higher scores indicated better health related quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Dave Burnett, Ph.D., Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No